CLINICAL TRIAL: NCT01507948
Title: The Neurobiology of Psychotherapy: Emotional Reactivity and Regulation in PTSD
Brief Title: Brain Imaging of Psychotherapy for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amit Etkin, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-10252011-8566
Record Dates: First submitted 2011-12-14; First posted 2012-01-11 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2015-07

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder (PTSD); Psychotherapy; non-medication treatment; Prolonged Exposure; Transcranial Magnetic Stimulation (TMS); Anxiety Disorders; emotion; emotion regulation; functional MRI; Affective Symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Emotional Regulation; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Prolonged Exposure Treatment (Experimental): Intake procedures include clinician-administered diagnostic battery, cognitive testing, self-report measures of symptoms, and functional imaging scan. Participants in this arm will complete a concurrent TMS/fMRI scan before beginning Prolonged Exposure (PE). PE will be delivered in 9-12 90-minute sessions. Therapy will be delivered by PhD-level therapists at Stanford and Palo Alto VA.
  Interventions: Behavioral: Prolonged exposure
- Wait list, immediately followed by Prolonged Exposure (No Intervention): Intake procedures include clinician-administered diagnostic battery, cognitive testing, self-report measures of symptoms, and functional imaging scan. NOTE: Participants in this arm receive treatment following a waitlist period of 12 weeks. After waitlist, will have a TMS/fMRI scan and then immediately begin Prolonged Exposure treatment. See above for description of Prolonged Exposure.

INTERVENTIONS:
Behavioral: Prolonged exposure — PE will be delivered in 9-12 90-minute sessions. Therapy will be delivered by PhD-level therapists at Stanford and Palo Alto VA. PE consists of four components: psychoeducation about PTSD symptoms and the behavioral or cognitive factors maintaining it, a brief breathing retraining that can be used as a stress management tool, prolonged imaginal exposure to the trauma memory both within-session and repeated as homework, and prolonged in vivo exposure to avoided scenarios in patients' day-to-day lives.
  Arms: Immediate Prolonged Exposure Treatment

SUMMARY:
The investigators are seeking people who have been exposed to a traumatic event in the past and have symptoms of posttraumatic stress disorder (PTSD) currently. A person with PTSD may feel significant distress when reminded of a traumatic event or feel depressed, anxious or jumpy.

As a part of this study, participants will receive brain MRIs and office assessments before and after psychotherapy. The investigators provide the gold-standard psychotherapy for PTSD, "Prolonged Exposure", free of charge; additionally participants are compensated for their time during assessment procedures. This study is exploring the brain circuitry involved in improvement in response to psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 60 years;
2. fMRI scanning eligibility, including no evidence of any form of metal embedded in the body (e.g., metal wires, nuts, bolts, screws, plates, sutures), as these produce artifacts when brain imaging;
3. not currently involved in an exposure-based psychotherapy, in order to be able to measure and interpret the effects of PE on PTSD;
4. must comprehend English well and show non-impaired intellectual abilities to ensure adequate comprehension of the fMRI task instructions and PE treatment;
5. no history of neurological or cardiovascular disorders, brain surgery, electroconvulsive or radiation treatment, brain hemorrhage or tumor, stroke, seizures or epilepsy, diabetes, hypo- or hyperthyroidism, head trauma with loss of consciousness greater than thirty minutes;
6. no regular use of benzodiazepine, opiate, thyroid, anticonvulsant or antipsychotic medications. Patients on stable doses of antidepressant medications will be allowed. Patients for whom antidepressant dosing is being actively titrated will be required to be on a stable dose for 1 month prior to inclusion in the study.

Exclusion Criteria:

* Any contraindication to being scanned in the 3T or 1.5T scanners at the Lucas Center or CNI such as having a pacemaker or implanted device that has not been cleared for scanning at the Lucas Center or CNI.
* Participants will be excluded from the study if there is any lifetime evidence of psychosis, mania, hypomania, or bipolar disorders. Other axis I comorbidities will not be a cause for exclusion.

In addition, subjects will be excluded if they have a significant CNS neurological condition such as stroke, seizure, tumor, hemorrhage, multiple sclerosis, etc.

Patients who have current substance dependence will be excluded from the study. A recent diagnosis of substance abuse is allowable, however, as long as subjects have been abstinent for greater than three months.

* Subjects will be excluded if they are currently in an exposure-based psychotherapy for PTSD.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2010-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD scale (CAPS) | Before and after Prolonged Exposure Treatment, which is expected to take approximately six weeks.
  The CAPS is a 30-item structured interview that corresponds to the DSM-IV criteria for PTSD. In addition to assessing the 17 PTSD symptoms, questions target the impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and frequency and intensity of five associated symptoms (guilt over acts, survivor guilt, gaps in awareness, depersonalization, and derealization). For each item, standardized questions and probes are provided.

SECONDARY OUTCOMES:
Mood and Anxiety Symptom Questionnaire (MASQ) | Before and after Prolonged Exposure Treatment, which is expected to take approximately six weeks.
  Treatment success based on Improvement on subscales of the MASQ, including decreased anxious arousal and decreased anhedonic depression, from pre- to post-treatment assessment
fMRI-assessed resting connectivity | Before and after Prolonged Exposure Treatment, which is expected to take approximately six weeks.
  From pre- to post-treatment, improve will be based on enhanced functional connectivity
Implicit emotion regulation | Assessed 4 times: Before beginning Prolonged Exposure, after the third week of therapy, after the last therapy session (on average 6 weeks after beginning therapy), and 1 month after the end of therapy.
  Implicit emotion regulation assessed through emotion conflict task performed during functional imaging. Performance based on reaction time and recruitment of emotion regulation regions during the task.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Etkin, M.D., Ph.D., Principal Investigator — Stanford University; Madeleine S Goodkind, Ph.D., Study Director — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Stanford University, Department of Psychiatry, Stanford, California

REFERENCES:
- [Derived] Fonzo GA, Goodkind MS, Oathes DJ, Zaiko YV, Harvey M, Peng KK, Weiss ME, Thompson AL, Zack SE, Lindley SE, Arnow BA, Jo B, Gross JJ, Rothbaum BO, Etkin A. PTSD Psychotherapy Outcome Predicted by Brain Activation During Emotional Reactivity and Regulation. Am J Psychiatry. 2017 Dec 1;174(12):1163-1174. doi: 10.1176/appi.ajp.2017.16091072. Epub 2017 Jul 18. PMID 28715908
- [Derived] Fonzo GA, Goodkind MS, Oathes DJ, Zaiko YV, Harvey M, Peng KK, Weiss ME, Thompson AL, Zack SE, Mills-Finnerty CE, Rosenberg BM, Edelstein R, Wright RN, Kole CA, Lindley SE, Arnow BA, Jo B, Gross JJ, Rothbaum BO, Etkin A. Selective Effects of Psychotherapy on Frontopolar Cortical Function in PTSD. Am J Psychiatry. 2017 Dec 1;174(12):1175-1184. doi: 10.1176/appi.ajp.2017.16091073. Epub 2017 Jul 18. PMID 28715907